CLINICAL TRIAL: NCT00959205
Title: Phase Ⅳ Study of CARTO 3D Mapping System vs Conventional Method in AF & VT
Brief Title: The Efficacy and Safety of CARTO 3D Mapping System Versus Conventional Method in AF and VT
Acronym: CARTOAF&VT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Korea University (Other)
Responsible Party: Young-Hoon Kim, Korea medical center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009_KU_CARTO
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2009-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Angiography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Angiography (Active Comparator): Conventional fluoroscopically guided activation mapping
  Interventions: Device: Angiography
- CARTO 3D (Experimental): CARTO (3D Electroanatomic imaging)
  Interventions: Device: CARTO 3D

INTERVENTIONS:
Device: CARTO 3D — CARTO (3D Electroanatomic imaging)
  Arms: CARTO 3D
Device: Angiography — Conventional fluoroscopically guided activation mapping
  Other Names: Celsius
  Arms: Angiography

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of electroanatomic imaging compared to conventional method in patients with VT.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of electroanatomic imaging (CARTO) compared to conventional fluoroscopically guided activation mapping (Conventional) method in patients with Atrial Fibrillation and Substrate-dependent Ventricular Tachycardia To evaluate cost-effectiveness of CARTO 3D image system compared to conventional method in the same study subjects

ELIGIBILITY:
Inclusion Criteria:

* patients with AF or substrate-dependent VT

Exclusion Criteria:

* administering with anticoagulants

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-06 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Fluoroscopic time | 24weeks
  Total duration of procedure using fluoroscopy on , in minute
Procedural duration | 24weeks
  Time from after puncture to catheter remover

SECONDARY OUTCOMES:
Ablation time | 24weeks
  Time from to Ablation
Procedural Success | 24weeks
  Achievement of the procedure endpoint for each arrhythmia
Clinical Success | 24weeks
  * 3 months freedom from recurrence of target arrhythmia
  * > 6 months freedom from recurrence of target arrhythmia
Radiation dose | 24weeks
  Calculated dose (in Gray) to the patient as recorded in the laboratory log
Morphology of ablation | 24weeks
  Number of Gap and the distance from the ostia of the pulmonary veins (In conventional group)
Complications | 24weeks
  * procedure and device related adverse event requiring any intervention to prevent permanent medical intervention
  * Important complications are reported individually
Cost Effectiveness | 24weeks
Survival Rate | 24weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kim Young-Hoon, MD, PhD, Principal Investigator — Korea medical center
Locations (5):
- South Korea (5):
  - Korea medical center, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Hospital/Internal Medicine, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Severance Hospital, Seoul